CLINICAL TRIAL: NCT05110261
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of Nirsevimab, a Monoclonal Antibody With Extended Half-life Against Respiratory Syncytial Virus, in Healthy Preterm and Term Infants in China
Brief Title: Evaluate the Safety and Efficacy of Nirsevimab in Healthy Preterm and Term Infants in China
Acronym: CHIMES
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: IQVIA RDS Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D5290C00006; 2021-005075-38 (EudraCT Number)
Record Dates: First submitted 2021-10-07; First posted 2021-11-05 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Lower Respiratory Tract Infection
Keywords: Respiratory Syncytial Viral (RSV); Efficacy; Safety; Nirsevimab; healthy Chinese preterm and term infants
MeSH Terms: interventions — nirsevimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nirsevimab (Experimental): Subjects will be randomized 2:1 to receive a single IM dose of nirsevimab or placebo.
  Interventions: Drug: Nirsevimab
- Placebo (Placebo Comparator): Subjects will be randomized 2:1 to receive a single IM dose of nirsevimab or placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nirsevimab — Drug: injection, 100 mg/mL, a single fixed IM dose of 50 mg (if weight < 5 kg) or 100 mg (if weight ≥ 5 kg)on day 1 only.
  Other Names: MEDI8897
  Arms: Nirsevimab
Drug: Placebo — Commercially available 0.9% (w/v) saline (sterile for human use) fixed IM dose of 0.5 mL (if weight <5 kg) or 1.0 mL (if weight >=5 kg)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the Safety and Efficacy of Nirsevimab, in Healthy Preterm and Term Infants in China

DETAILED DESCRIPTION:
This is a Phase 3 randomized, double-blind, placebo-controlled, single-dose study to determine if nirsevimab will prevent medically attended RSV-confirmed LRTI in healthy preterm and term infants entering their first RSV season. The population to be enrolled is healthy preterm and term infants > 29 weeks 0 days GA entering their first RSV season, who would not receive RSV prophylaxis based on the American Academy of Pediatrics (AAP) or other local or national guidelines. Approximately 800 subjects will be randomized 2:1 to receive a single IM dose of nirsevimab 50 mg (if weight < 5 kg) or 100 mg (if weight ≥ 5 kg) (N = 530) or placebo (N = 270). Randomization will be stratified by subject age at the time of randomization (≤ 3 months, > 3 to ≤ 6 months, > 6 months), and by GA (< 35 weeks GA, ≥ 35 weeks GA). Enrollment of infants > 6 months of age will be limited to approximately 100. All subjects will be followed through 1 year after dose administration. An independent data monitoring committee will review safety data regularly and make recommendations regarding further study conduct. Around 40 investigational study centres participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese preterm and term infants in their first year of life and born ≥ 29 weeks 0 days GA (infants who have an underlying illness such as cystic fibrosis or Down syndrome with no other risk factors are eligible)
2. Infants who are entering their first RSV season at the time of screening
3. Written informed consent and any locally required authorization obtained from the subject's parent(s)/legal representative(s) prior to performing any protocol-related procedures, including screening evaluations
4. Subject's parent(s)/legal representative(s) able to understand and comply with the requirements of the protocol including follow-up visits as judged by the Investigator
5. Subject is available to complete the follow up period, which will be approximately 1 year after receipt of investigational product

Exclusion Criteria:

1. Any fever (≥ 100.4°F [≥ 38.0°C], regardless of route) or acute illness within 7 days prior to investigational product administration
2. Any history of LRTI or active LRTI prior to, or at the time of, randomization
3. Known history of RSV infection or active RSV infection prior to, or at the time of, randomization
4. Any drug therapy (chronic or other) within 7 days prior to randomization or expected receipt during the study with the exception of: a) multivitamins and iron; b) infrequent use of over-the-counter (OTC) medications for the systemic treatment of common childhood symptoms (eg, pain relievers) that may be permitted according to the judgment of the Investigator
5. Any current or expected receipt of immunosuppressive agents including steroids (except for the use of topical steroids according to the judgment of the Investigator)
6. History of receipt of blood products, or immunoglobulin products, or expected receipt through the duration of the study
7. Hospitalization at the time of randomization, unless discharge is expected within the 7 days after randomization
8. Known renal impairment
9. Known hepatic dysfunction including known or suspected active or chronic hepatitis infection
10. History of CLD/bronchopulmonary dysplasia
11. Clinically significant congenital anomaly of the respiratory tract
12. CHD, except for children with uncomplicated CHD (eg, patent ductus arteriosus, small septal defect)
13. Chronic seizure, or evolving or unstable neurologic disorder
14. Prior history of a suspected or actual acute life-threatening event
15. Known immunodeficiency, including human immunodeficiency virus (HIV)
16. Mother with HIV infection (unless the child has been proven to be not infected)
17. Any known allergy or history of allergic reaction to immunoglobulin products, blood products, or other foreign proteins, or history of allergic reaction
18. Receipt of palivizumab or other RSV mAb or any RSV vaccine, including maternal RSV vaccination
19. Receipt of any monoclonal or polyclonal antibody (for example, hepatitis B immune globulin, IV immunoglobulin) or anticipated use during the study
20. Receipt of any investigational product
21. Concurrent enrollment in another interventional study
22. Any condition that, in the opinion of the Investigator, would interfere with evaluation of the investigational product or interpretation of study results
23. Children of employees of the Sponsor, clinical study site, or any other individuals involved with the conduct of the study, or immediate family members of such individuals

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2025-11-24 (Estimated); Study Completion 2025-11-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of medically attended LRTI due to RT-PCR-confirmed RSV | Day 1 to Day 151
  The incidence of medically attended RSV LRTI (inpatient and outpatient) through 150 days post dose (ie, during a typical 5-month RSV season) for all infants, based on RSV test results (performed centrally using RT-PCR) and objective protocol-defined LRTI criteria, is the primary endpoint and will be presented by treatment groups. For subjects with multiple events, only the first occurrence will be used in the analysis. RSV LRTI that occurs through 150 days post dose will contribute to the primary efficacy analysis.

SECONDARY OUTCOMES:
Incidence of RSV Hospitalization RT PCR-confirmed RSV | Day 1 to Day 151
  To assess the efficacy of nirsevimab in reducing hospitalizations due to protocol-defined LRTI caused by RT-PCR-confirmed RSV, compared to placebo
Safety and tolerability | Day 1 to Day 361
  Safety and tolerability of Nirsevimab as assessed by the occurrence of all treatment emergent adverse events (TEAEs) and treatment emergent serious adverse events (TESAE) Safety of Nirsevimab will primarily be assessed and measured by the occurrence of all treatment-emergent AEs and SAEs.
  Other safety assessments will include the occurrence of Adverse Event of Special Interest (AESIs) and New Onset Chronic Diseases (NOCDs).
Summary of nirsevimab serum concentrations | Day 1, Day 15, Day 151 & Day 361
  To evaluate serum concentrations of nirsevimab.
Incidence of ADA to nirsevimab in serum | Day 1, Day 151 & Day 361
  To evaluate ADA responses to nirsevimab in serum.

CONTACTS AND LOCATIONS:
Locations (26):
- China (26):
  - Research Site, Beijing
  - Research Site, Changde
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Jiaxing
  - Research Site, Kunming
  - Research Site, Langfang
  - Research Site, Linfen
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Sanmenxia
  - Research Site, Sanya
  - Research Site, Shantou
  - Research Site, Shaoxing
  - Research Site, Shenzhen
  - Research Site, Suzhou
  - Research Site, Tangshan
  - Research Site, Tianjin
  - Research Site, Tonghua
  - Research Site, Wenzhou
  - Research Site, Wuxi
  - Research Site, Xinxiang
  - Research Site, Zhengzhou
  - Research Site, Zhongshan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home